CLINICAL TRIAL: NCT05233176
Title: Kinetics of C-Reactive Protein During the Overall Management of Acute Coronary Syndrome Treated by Transluminal Angioplasty
Brief Title: Kinetics of C-Reactive Protein During the Management of Acute Coronary Syndrome Treated by Transluminal Angioplasty
Acronym: CRP KIN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP 211274; 2021-A02081-40 (Other: IDRCB)
Record Dates: First submitted 2022-01-28; First posted 2022-02-10 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; C reactive protein; kinetic; adults
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — C reactive protein (CRP) sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objective of the study focuses on the kinetics of plasma CRP measured during the overall management (before the angioplasty procedure until the discharge of hospitalization) of patients with ST+ ACS requiring emergency transluminal angioplasty.

DETAILED DESCRIPTION:
During the management of acute coronary syndrome with ST segment elevation (ACS-ST+), an ischemia-reperfusion syndrome is observed in connection with primary coronary occlusion (ischemia) and percutaneous angioplasty during the therapeutic coronary reperfusion.

This ischemia-reperfusion syndrome results biologically in an inflammatory syndrome evaluated in particular by the assay of C-reactive protein (CRP). CRP is a marker of inflammation used in routine practice. Previous studies have reported the prognostic value of CRP at the 48th hour of hospital treatment for ST+ ACS. If the value of CRP is correlated with the risk of mortality and heart failure, the fact remains that no study has, to date, studied its kinetics during the overall management (pre and intra-hospital) of ACS ST+. This is all the more important since the previous therapies taken by the patient (statins for example) and/or those administered during treatment (colchicine, ticagrelor, anti-GPIIbIIIa are capable of modifying the pre-hospital value of the CRP.

In this study, the kinetics of plasma CRP measured during the first medical contact (emergency, cardiology or resuscitation), then, in the catheterization room before the angioplasty procedure, then in the catheterization room, after the angioplasty, then at the 6th hour (H6), at the 12th hour (H12), at the 24th hour (H24), at the 48th hour (H48) and once a week until the 7th day then once a week until discharge hospitalization with a maximum of 30 days of follow-up, as part of the usual follow-up of patients with ST+ ACS requiring emergency transluminal angioplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old;
* ST+ ACS requiring emergency transluminal angioplasty;
* Affiliation to a social security scheme or beneficiary.

Exclusion Criteria:

* ST+ ACS not requiring emergency transluminal angioplasty;
* Pregnancy;
* Under guardianship or curatorship;
* Foreign patient under french AME scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients cared for ST+ ACS requiring emergency transluminal angioplasty.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Plasma CRP kinetic | Pre-angioplasty, hour 6, hour 12, hour 24, hour 48 and daily post angioplasty until day 7 then weekly untill day 30
  Blood sampling: Pre-angioplasty, on H6, H12, H24, H48 and once a day post angioplasty until the 7th day; then once a week until discharge from hospital with a maximum of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Romain Jouffroy, MD, PhD, Principal Investigator — Intensive Care Unit - Ambroise Paré Hospital - APHP; Marie Hauguel-Moreau, MD, Study Director — Cardiology department, Ambroise Paré hospital, APHP
Locations (2):
- France (2):
  - Cardiology department, Ambroise Paré hospital, APHP, Boulogne-Billancourt
  - Intensive care unit, Ambroise Paré hospital, APHP, Boulogne-Billancourt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milwidsky A, Ziv-Baran T, Letourneau-Shesaf S, Keren G, Taieb P, Berliner S, Shacham Y. CRP velocity and short-term mortality in ST segment elevation myocardial infarction. Biomarkers. 2017 May-Jun;22(3-4):383-386. doi: 10.1080/1354750X.2017.1279218. Epub 2017 Jan 25. PMID 28055283